CLINICAL TRIAL: NCT04945213
Title: Biperiden for Prevention of Epilepsy in Patients With Traumatic Brain Injury
Brief Title: Biperiden Trial for Epilepsy Prevention
Acronym: BIPERIDEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: PROADI-SUS (Unknown); Ministry of Health, Brazil (Other Government); University of Sao Paulo (Other); Santa Casa de Campo Grande (Other); Hospital Sao Rafael (Other); Santa Casa de Misericórdia de Sobral (Unknown); Hospital de Clinicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (Unknown); Hospital São Paulo, Universidade Federal de São Paulo (Unknown); Instituto Doutor José Frota (Unknown); Hospital São Vicente de Paulo (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AVAP-NG 1983; 39005920810015461 (Other: Ethics Board of Sirio-Libanês Hospital)
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-11

CONDITIONS: Brain Injury Traumatic Moderate; Brain Injury Traumatic Severe; Post Traumatic Epilepsy
Keywords: Brain Injury; Epilepsy; Biperiden
MeSH Terms: conditions — Epilepsy, Post-Traumatic; Brain Injuries; Epilepsy | interventions — Biperiden; Sodium Lactate; Lactic Acid; Sodium Hydroxide; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biperiden (Experimental): Drug: Biperiden 5mg of biperiden diluted in 100 ml of 0.9% saline - every 6 hours for 10 consecutive days - IV
  Interventions: Drug: Biperiden
- Placebo (Placebo Comparator): Placebo
  1 mL of sterile vehicle (sodium lactate, lactic acid, sodium hydroxide and water for injections) diluted in 100 mL of 0,9% saline - every 6 hours for 10 consecutive days - IV
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Biperiden — 5mg of biperiden diluted in 100 ml of 0.9% saline - every 6 hours for 10 consecutive days - IV
  Other Names: Akineton
  Arms: Biperiden
Other: Placebo — 1ml sterile vehicle (sodium lactate, lactic acid, sodium hydroxide and water for injections) diluted in 100 ml 0.9% saline - every 6 hours for 10 consecutive days - IV
  Other Names: Sterile vehicle (sodium lactate, lactic acid, sodium hydroxide and water for injections)
  Arms: Placebo

SUMMARY:
One of the most important neurological consequences following Traumatic Brain Injury (TBI) is the development of post traumatic epilepsy (PTE). Nevertheless, there is still no effective therapeutic intervention to reduce the occurrence of PTE. In previous studies with animals models of epilepsy, the biperiden decreased the incidence and intensity of spontaneous epileptic seizures besides delaying their appearance. The aim of this study is the evaluation of biperiden as antiepileptogenic drug to prevent PTE and also the determination of side effects, evaluating its cost-effectiveness in patients with moderate and severe TBI.

DETAILED DESCRIPTION:
One of the most important neurological consequences following Traumatic Brain Injury (TBI) is the development of post traumatic epilepsy (PTE), which accounts for 5% of all epilepsy etiologies in the general population. This makes TBI one of the most important causes of secondary epilepsy, overcoming other causes such as infections, drug abuse or familiar history of epilepsy. The occurrence of spontaneous epileptic seizures after TBI, mostly starting in the first 2 years after moderate or severe TBI, might be as high as 86%, specially in those with a single acute symptomatic seizure, with remission rates of 25-40%. The causative relationship between TBI and epilepsy, as well as other types of epilepsy in general, are still not completely understood and PTE is not yet preventable.

The therapeutic approach indicated for TBI may involve medications, surgical procedures or both, with no effective therapeutic intervention to reduce its occurrence. Several experimental studies in animal models have shown that drugs, which modify processes of neuronal plasticity, have the potential to modify the natural course of PTE. Among these, biperiden (anti-cholinergic indicated for Parkinson's disease) has shown reduction in the incidence and intensity of spontaneous epileptic seizures and also delayed their occurence in animal epilepsy model. Thus Biperiden would be an excellent candidate for an antiepileptogenic agent. It is intended here to test its effectiveness and safety in adult patients, victims of moderate and severe TBI. Patients will be randomized to receive 5 mg of Biperiden iv, diluted in 100 ml of 0.9% saline (treatment group) or 1 mL of sterile vehicle (sodium lactate, lactic acid, sodium hydroxide and water for injections) diluted in 100 mL of 0,9% saline (placebo group), every 6 hours for 10 days after TBI. Prospectively, patients will be followed up for two years, on periodic visits to assess the development of epileptic seizures. Other factors that might have benefits with the treatment, such as epileptiform abnormalities, genetic markers and neuropsychological aspects, will also be evaluated. The results could be important for a better comprehension of basic mechanisms of epilepsy development. Side effects of Biperiden use, at high doses during a short period of time, will be measured. If Biperiden is efficient and safe, it will certainly be a low-cost option for Brazilian public health system (SUS).

ELIGIBILITY:
Inclusion Criteria:

* Given informed consent
* 18 - 75 years of age
* GCS between 6 and 12 at hospital admission. GCS between 3 and 5 at hospital admission can be enrolled if patient was sedated at the accident scene with previous GCS between 6 and 15.
* Moderate or severe acute traumatic brain injury
* All genders
* Brain CT scan with signs of of acute intraparenchymal hemorrhage and/or contusion
* Able to receive the first dose of treatment or placebo within 18 hours of brain injury,

Exclusion Criteria:

* Previous use of biperiden
* History of epilepsy (confirmed by patient chart)
* History of seizures or use of antiepileptic medication
* Pregnancy
* Participation in another clinical trial at the time of randomization
* History of neoplasia, neurodegenerative diseases; history of stroke, cognitive impairment, benign prostatic hyperplasia, atrioventricular block or any other cardiac arrhythmia, or glaucoma megacolon or mechanical obstruction
* Homeless patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post Traumatic Epilepsy (PTE) | 7 days to 24 months
  Participants who present epileptic seizures will be compared between placebo and biperiden groups. Seizures will be counted starting 7 days after TBI and continuously during the following two years follow-up period. Patients and their relatives will be asked to keep a diary of seizures, and record all seizures with detailed descriptions of each event.
Occurrence of Severe Adverse Events | 24 months
  Proportion of participants that present at least one severe adverse event until 24 months after the traumatic brain injury will be compared between biperiden and placebo groups.

SECONDARY OUTCOMES:
Electroencephalogram Analyses: Presence of Epileptiform Discharges | 1,3, 6, 9,12,18 and 24 months
  Electroencephalogram (EEG) will be analysed mostly looking for epileptiform abnormalities and ictal patterns. EEG is going to be recorded at follow-up visits. Data will be compared between placebo and biperiden groups.
Neuropsychological Assessments - semantic memory | 6 and 24 months
  Standard neuropsychologic test (Vocabulary) of the Wechsler Intelligence Scale III (WAIS III) which will be applied by psychologists at 6 months and then 24 months after TBI. It evaluate the semantic memory. It will be used the percentile scale that varies between 0.1 minimum (worst result) and 99.9 maximum (best result). The results will be compared between biperiden and placebo groups.
Neuropsychological Assessments - visual construction | 6 and 24 months
  Standard neuropsychologic test (Block design) of the Wechsler Intelligence Scale III (WAIS III) which will be applied by psychologists at 6 months and then 24 months after TBI. It evaluates the visual construction. It will be used the percentile scale that varies between 0.1 minimum (worst result) and 99.9 maximum (best result). The results will be compared between biperiden and placebo groups.
Neuropsychological Assessments - information processing speed and attention | 6 and 24 months
  Standard neuropsychologic test (Digit Symbol-Coding and Symbol Search) of the Wechsler Intelligence Scale III (WAIS III) which will be applied by psychologists at 6 months and then 24 months after TBI. It evaluates the information processing speed and attention. It will be used the percentile scale that varies between 0.1 minimum (worst result) and 99.9 maximum (best result). The results will be compared between biperiden and placebo groups.
Neuropsychological Assessments - short term memory | 6 and 24 months
  Standard neuropsychologic test (Digit Span) of the Wechsler Intelligence Scale III (WAIS III) which will be applied by psychologists at 6 months and then 24 months after TBI. It evaluates the information processing speed and attention. It will be used the percentile scale that varies between 0.1 minimum (worst result) and 99.9 maximum (best result). The results will be compared between biperiden and placebo groups.
Neuropsychological Assessments - visual construction and visuospatial long-term memory | 6 and 24 months
  Standard neuropsychologic test (Rey-Osterrieth complex figure) which will be applied by psychologists at 6 months and then 24 months after TBI. It evaluates the visual construction and visuospatial long-term memory. It will be used the percentile scale that varies between 0.1 minimum (worst result) and 99.9 maximum (best result). The results will be compared between biperiden and placebo groups.
Neuropsychological Assessments - verbal long-term memory | 6 and 24 months
  Standard neuropsychologic test (Rey Auditory Verbal Learning Test (RAVLT)) which will be applied by psychologists at 6 months and then 24 months after TBI. It evaluates the verbal long-term memory. It will be used the percentile scale that varies between 0.1 minimum (worst result) and 99.9 maximum (best result). The results will be compared between biperiden and placebo groups.
Neuropsychological Assessments - executive functions | 6 and 24 months
  Standard neuropsychologic test (Five Digit Test (FDT)) which will be applied by psychologists at 6 months and then 24 months after TBI. It evaluates the verbal long-term memory. It will be used the percentile scale that varies between 0.1 minimum (worst result) and 99.9 maximum (best result). The results will be compared between biperiden and placebo groups.
Health-related quality of life assessment - EQ-5D-3L descriptive system | 3, 6, 12 and 24 months
  Health related quality of life will be evaluated through the portuguese version of EuroQol three-level version (EQ-5D-3L) descriptive system. EQ-5D-3L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state in each of the five dimensions. The answers given to ED-5D-3L can be converted into EQ-5D index, an utility scores anchored at - 0,78 for the worst health to 1 for perfect health. Results will be compared between biperiden and placebo groups.
Health-related quality of life assessment - EQ-VAS self-rated health | 3, 6, 12 and 24 months
  Health related quality of life will be evaluated through the portuguese version of EuroQol visual analogue scale (EQ-VAS) which records the patient's self-rated health on a vertical visual analogue scale and it can be used as a quantitative measure of health outcome that reflects the patient's own judgement. EQ-VAS has a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status). Results will be compared between biperiden and placebo groups.
Biomarkers - Expression of the ApoEϵ4 allele [ Time Frame: 10 days after TBI ] | Up to 10 days after TBI
  To investigate the expression of the ApoEϵ4 allele in TBI patients, its correlation with post traumatic epilepsy and the biperiden response to prevent epilepsy, RFLP-PCR will be assayed in blood samples of TBI patients. The genotyping reactions will be performed blinded to clinical data. The presence of the ApoEϵ4 allele will be correlated with the incidence of seizures in the follow-up assessments after TBI.
Incidence of Post Traumatic Epilepsy (PTE) during the Follow-up | 1,3, 6, 9,12,18 and 24 months
  Participants who present epileptic seizures will be compared between placebo and biperiden groups. Seizures will be counted starting 7 days after TBI and continuously during the following two years follow-up period. For each visit after TBI patients and their relatives will be asked about occurrence of seizures and their diary notes of seizures. For all events, a detailed descriptions wiil be asked . Seizures should be classified according to 2017 International League against Epilepsy classification. The recordings will be evaluated in each patient visit. The goal is to define, over time, when epilepsy starts in each group (biperiden and placebo).

OTHER OUTCOMES:
Incidence of Mortality | 24 months
  Participants who died throughout the period of study (24 months after TBI) will be compared between placebo and biperiden groups. Although patients includes are severe, the effectiveness of biperiden to reduce mortality might be evaluated,
Incidence of Non-Severe Adverse Events | 1,3, 6, 9,12,18 and 24 months
  Biperiden and placebo groups will be compared for occurrence of any non-severe adverse events at each visit of follow-up, from 1 month to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz E Mello, MD, PhD, Principal Investigator — Hospital Sirio-Libanês; Eliana Garzon, MD, PhD, Principal Investigator — Hospital Sirio-Libanês
Locations (10):
- Brazil (10):
  - Instituto Doutor José Frota, Fortaleza, Ceará
  - Santa Casa de Misericórdia de Sobral, Sobral, Ceará
  - Hospital Estadual Urgencia e Emergencia -HEUE, Vitória, Espírito Santo
  - Hospital São Rafael, Salvador, Estado de Bahia
  - Associação Beneficente Santa Casa de Campo Grande, Campo Grande, Mato Grosso do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Hospital Sirio-Libanes, São Paulo
  - Hospital São Paulo, Universidade Federal de São Paulo, São Paulo

REFERENCES:
- [Background] Antoniuk SA. [Non-epileptic disorders in infancy and adolescence]. Medicina (B Aires). 2013;73 Suppl 1:71-6. Spanish. PMID 24072054
- [Background] Annegers JF, Hauser WA, Coan SP, Rocca WA. A population-based study of seizures after traumatic brain injuries. N Engl J Med. 1998 Jan 1;338(1):20-4. doi: 10.1056/NEJM199801013380104. PMID 9414327
- [Background] Aronstam, RS & Patil, P. Muscarinic Receptors: Autonomic Neurons, Encyclopedia of Neuroscience, Academic Press,2009; 1141-1149, ISBN 9780080450469, https://doi.org/10.1016/B978-008045046-9.00692-6.
- [Background] Anvisa. MANUAL PARA NOTIFICAÇÃO DE EVENTOS ADVERSOS E MONITORAMENTO DE SEGURANÇA EM ENSAIOS CLÍNICOS - 1a. edição. 2016. Disponível em: http://portal.anvisa.gov.br/documents/33836/2492465/Manual+para+Notifica%C3%A7%C3%A3o+de+Eventos+Adversos+e+Monitoramento+de+Seguran%C3%A7a+em+Ensaios+Cl%C3%ADnicos+-+1%C2%AA+Edi%C3%A7%C3%A3o/04a68574-8aac-43c9-b0b2-7b7cd80831c4. Acessado em 5 de novembro de 2019.
- [Background] Brady RD, Casillas-Espinosa PM, Agoston DV, Bertram EH, Kamnaksh A, Semple BD, Shultz SR. Modelling traumatic brain injury and posttraumatic epilepsy in rodents. Neurobiol Dis. 2019 Mar;123:8-19. doi: 10.1016/j.nbd.2018.08.007. Epub 2018 Aug 16. PMID 30121231
- [Background] Bittencourt S, Ferrazoli E, Valente MF, Romariz S, Janisset NRLL, Macedo CE, Antonio BB, Barros V, Mundim M, Porcionatto M, Aarao MC, Miranda MF, Rodrigues AM, de Almeida AG, Longo BM, Mello LE. Modification of the natural progression of epileptogenesis by means of biperiden in the pilocarpine model of epilepsy. Epilepsy Res. 2017 Dec;138:88-97. doi: 10.1016/j.eplepsyres.2017.10.019. Epub 2017 Oct 29. PMID 29096134
- [Background] D'Ambrosio R, Perucca E. Epilepsy after head injury. Curr Opin Neurol. 2004 Dec;17(6):731-5. doi: 10.1097/00019052-200412000-00014. PMID 15542983
- [Background] da Silva AM, Vaz AR, Ribeiro I, Melo AR, Nune B, Correia M. Controversies in posttraumatic epilepsy. Acta Neurochir Suppl (Wien). 1990;50:48-51. doi: 10.1007/978-3-7091-9104-0_9. PMID 2129092
- [Background] de Almeida CE, de Sousa Filho JL, Dourado JC, Gontijo PA, Dellaretti MA, Costa BS. Traumatic Brain Injury Epidemiology in Brazil. World Neurosurg. 2016 Mar;87:540-7. doi: 10.1016/j.wneu.2015.10.020. Epub 2015 Oct 17. PMID 26485419
- [Background] DeVito NJ, Goldacre B. Catalogue of bias: publication bias. BMJ Evid Based Med. 2019 Apr;24(2):53-54. doi: 10.1136/bmjebm-2018-111107. Epub 2018 Dec 6. No abstract available. PMID 30523135
- [Background] Englander J, Bushnik T, Duong TT, Cifu DX, Zafonte R, Wright J, Hughes R, Bergman W. Analyzing risk factors for late posttraumatic seizures: a prospective, multicenter investigation. Arch Phys Med Rehabil. 2003 Mar;84(3):365-73. doi: 10.1053/apmr.2003.50022. PMID 12638104
- [Background] Husereau D, Drummond M, Petrou S, Carswell C, Moher D, Greenberg D, Augustovski F, Briggs AH, Mauskopf J, Loder E; CHEERS Task Force. Consolidated Health Economic Evaluation Reporting Standards (CHEERS) statement. Value Health. 2013 Mar-Apr;16(2):e1-5. doi: 10.1016/j.jval.2013.02.010. PMID 23538200
- [Background] Benassi SK, Alves JGSM, Guidoreni CG, Massant CG, Queiroz CM, Garrido-Sanabria E, Loduca RDS, Susemihl MA, Paiva WS, de Andrade AF, Teixeira MJ, Andrade JQ, Garzon E, Foresti ML, Mello LE. Two decades of research towards a potential first anti-epileptic drug. Seizure. 2021 Aug;90:99-109. doi: 10.1016/j.seizure.2021.02.031. Epub 2021 Mar 3. PMID 33714677
- [Background] Hauser WA, Annegers JF, Kurland LT. Prevalence of epilepsy in Rochester, Minnesota: 1940-1980. Epilepsia. 1991 Jul-Aug;32(4):429-45. doi: 10.1111/j.1528-1157.1991.tb04675.x. PMID 1868801
- [Derived] Foresti ML, Garzon E, Pinheiro CCG, Pacheco RL, Riera R, Mello LE. Biperiden for prevention of post-traumatic epilepsy: A protocol of a double-blinded placebo-controlled randomized clinical trial (BIPERIDEN trial). PLoS One. 2022 Sep 9;17(9):e0273584. doi: 10.1371/journal.pone.0273584. eCollection 2022. PMID 36084082